CLINICAL TRIAL: NCT00734903
Title: A Randomized Controlled Trial on Women's Substance Abuse Treatment
Brief Title: Women Veterans' Substance Abuse Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEUA-001-08S
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-02

CONDITIONS: Substance Use Disorders
Keywords: Women; Substance Use Disorders; Treatment Efficacy; Women's Health; Outcome Assessment (Health Care)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Woman's Path to Recovery (WPR) (Experimental): A gender-focused approach to addiction recovery
  Interventions: Behavioral: A Woman's Path to Recovery
- 12-Step Facilitation (TSF) (Active Comparator): An evidence-based, non-gender-focused approach to addiction recovery
  Interventions: Behavioral: 12-Step Facilitation

INTERVENTIONS:
Behavioral: A Woman's Path to Recovery — WPR is a gender-specific therapy model for women with substance use disorder. It uses A Woman's Addiction Workbook to provide education and coping skills. In this trial it was conducted in 12 weekly individual sessions.
  Other Names: A Woman's Addiction Workbook
  Arms: A Woman's Path to Recovery (WPR)
Behavioral: 12-Step Facilitation — 12SF is an evidence-based therapy designed to facilitate early recovery from substance addiction. It is an individual model consisting of 12 sessions that use the principles of 12-step groups such as Alcoholics Anonymous, and strongly emphasizes participation in those. In this trial the model was conducted weekly.
  Arms: 12-Step Facilitation (TSF)

SUMMARY:
The purpose of this study is to examine the efficacy of a gender-focused addiction treatment model (A Woman's Path to Recovery) versus a non-gender focused addiction treatment model (12-Step Facilitation) in a sample of women Veterans with substance use disorder.

DETAILED DESCRIPTION:
Substance use disorder (SUD) is problem among women military Veterans, especially younger ones. The goal of this study was to examine the efficacy a gender-focused model of SUD treatment (A Woman's Path to Recovery, WPR) compared to an evidence-based active comparator that is not gender-specific (12-Step Facilitation, 12SF), in a sample of for women Veterans. The investigators randomized 66 women Veterans, ages 18-65, who were diagnosed with current SUD and used substances in the last 90 days. The treatment phase was 12 weekly individual therapy sessions and all participants could also obtain treatment-as-usual (any other treatments they chose to attend). Assessments were conducted at baseline, end of treatment and 3-month follow up. Sample size was based on power analysis (an effect of .80 at a .05 level of significance). The primary outcome variable was substance use, with various secondary outcomes also studied (e.g., psychosocial functioning, psychiatric symptoms, coping skills, 12-step attendance). Urinalysis / breathalyzer (biological measures) were also included to validate substance use self-report. The investigators hypothesized that participants in the experimental condition (WPR) would have more positive outcomes on both primary and secondary variables compared to those in the comparison condition (12SF). The investigators also hypothesized that WPR patients would increase coping skills more and 12SF would increase 12-step attendance more, relative to the other condition.

ELIGIBILITY:
Inclusion Criteria:

* Female Veteran
* 18-65 years of age
* Meet DSM-IV criteria for current SUD with "current" defined as meeting SUD criteria per the DSM-IV and having used a substance within the 90 days prior to intake (to be able to accurately evaluate changes in their substance use from baseline)
* Plan to stay in the Boston area for the next 6 months
* Have a mailing address and live close enough to come to the hospital once weekly for treatment and/or assessment
* Able to complete the Statement of Informed Consent
* Willing to participate in all assessments and breathalyzer/urine testing
* Willing to provide a release of information such that study staff can contact her other providers as needed regarding any concerns during her participation
* Able to obtain medical clearance
* Willing to allow us to contact family and/or friends if participant loses contact with us
* Literate
* Not pregnant or planning to become pregnant

Exclusion Criteria:

* Any acute medical condition that would interfere with the participant's ability to participate in treatment, or would be of such severity as to affect the individual's psychological functioning (e.g., cancer)
* Current bipolar I disorder, schizophrenia or other psychotic disorders or mental retardation or organic mental disorder (determined by screening interview)
* Any clinical sign that the client is not sufficiently stable to participate in the treatment, such as client's treatment provider indicating that participation in the treatment would be contraindicated
* Dangerousness that would present a threat to other staff or other clients (e.g., history of recent assault)
* Client is mandated to treatment
* Psychopharmacologic treatment that is planned to change or likely to change substantively over the 3-month active treatment phase (with "substantive" defined as any addition of a new medication or major shift in dosage)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Najavits, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Najavits LM, Enggasser J, Brief D, Federman E. A randomized controlled trial of a gender-focused addiction model versus 12-step facilitation for women veterans. Am J Addict. 2018 Apr;27(3):210-216. doi: 10.1111/ajad.12709. PMID 29596724

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 103 screened, 82 were eligible, 21 ineligible. Of 82 eligible, 66 completed baseline and were randomized; 16 did not complete baseline.
Period: Overall Study
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Started | 33 | 33
Completed End of Treatment Assessment | 21 | 23
Completed 3-month Followup | 14 | 15
Completed (Completion was defined, a priori, as completing at least 2 study assessments) | 30 | 32
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF) | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.97 (9.92) | 48.45 (8.13) | 47.72 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 23 | 22 | 45
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Addiction Severity Index Alcohol Composite
Description: Alcohol use and associated problems as measured by blinded-interviewer rated composite score. Six questions comprise the alcohol composite, of which 4 are answered from 0-30 (number of days in past month) and 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome). Breathalyzer was also obtained to verify self-report and was coded as positive (worst pathology, means patient was intoxicated) or negative (not pathological; patient was not intoxicated).
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | .36 (.24) | .46 (.35)
  End of Treatment | .18 (.21) | .26 (.24)
  3-month followup | .23 (.19) | .21 (.11)

2. Primary Outcome: Addiction Severity Index Drug Composite
Description: Drug use and associated problems as measured by blinded-interviewer rated composite score. Urinalysis/breathalyzer is also obtained to verify self-report.Drug use and associated problems as measured by blinded-interviewer rated composite score. Eleven questions comprise the drug composite, of which 9 are answered from 0-30 (number of days in past month) and 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome). Urinanalysis was also obtained to verify self-report and was coded as positive (worst pathology, means patient was intoxicated) or negative (not pathological; patient was not intoxicated).
Time Frame: Baseline, end of treatment (3 months), and 3-month post-treatment followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | .10 (.11) | .10 (.12)
  End of Treatment | .04 (.05) | .06 (.06)
  3-month followup | .04 (.05) | .04 (.05)

3. Primary Outcome: Brief Addiction Monitor
Description: Assesses number of days in the past 30 days that person used substances including alcohol and drugs
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: days out of past 30 days
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 31 | 31
days out of past 30 days
  Baseline | 4.61 (3.50) | 4.48 (3.85)
  End of Treatment | 1.96 (2.08) | 2.33 (3.17)
  3-month followup | 2.33 (1.92) | 1.92 (2.36)

4. Secondary Outcome: Addiction Severity Index Medical Composite Score
Description: Medical problems associated with substance use as measured by blinded-interviewer rated composite score. Several questions are answered from 0-30 (number of days in past month) and the remaining 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome).
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 27 | 28
units on a scale
  Baseline | .38 (.31) | .43 (.38)
  End of Treatment | .38 (.29) | .33 (.30)
  3-month followup | .21 (.28) | .20 (.28)

5. Secondary Outcome: Addiction Severity Index Employment Composite
Description: Employment problems associated with substance use as measured by blinded-interviewer rated composite score. Several questions are answered from 0-30 (number of days in past month) and the remaining 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome).
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 27 | 28
units on a scale
  Baseline | .64 (.27) | .59 (.34)
  End of Treatment | .58 (.29) | .54 (.33)
  3-month followup | .58 (.28) | .56 (.32)

6. Secondary Outcome: Addiction Severity Index Psychiatric Composite
Description: Psychiatric problems associated with substance use as measured by blinded-interviewer rated composite score. Several questions are answered from 0-30 (number of days in past month) and the remaining 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome).
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 27 | 28
units on a scale
  Baseline | .43 (.21) | .48 (.18)
  End of Treatment | .37 (.21) | .41 (.18)
  3-month followup | .31 (.21) | .39 (.19)

7. Secondary Outcome: Addiction Severity Index Family/Social Composite
Description: Family/social problems associated with substance use as measured by blinded-interviewer rated composite score. Several questions are answered from 0-30 (number of days in past month) and the remaining 2 are subjective Likert ratings 0 (not at all) to 4 (extremely), with higher scores on all items indicating worse pathology. Composite scores are computed and range from 0 (worst outcome) to 1 (best outcome).
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | .20 (.21) | .29 (.22)
  End of Treatment | .14 (.15) | .22 (.29)
  3-month followup | .23 (.23) | .30 (.24)

8. Secondary Outcome: Global Severity Index of the Brief Symptom Inventory
Description: Self-report measure of severity of general psychiatric symptoms ranging from 0 (not at all) to 4 (extremely). The total scale score Global severity index (GSI) is the mean of all 53 items on the measures. The mean ranges from 0 to 4, with higher indicating worse pathology.
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 31 | 31
units on a scale
  Baseline | 1.55 (1.21) | 1.85 (1.12)
  End of Treatment | 1.37 (1.14) | 1.34 (.92)
  3-month followup | 1.62 (1.01) | 1.26 (.88)

9. Secondary Outcome: BASIS-24 Psychosocial Functioning
Description: 24 items that address how patients feel before and after receiving care. The survey measures the degree of difficulty experienced by the patient during a one-week period on a five-point scale ranging from 0 (no difficulty) to extreme difficulty (4) with the overall score ranging from 0-96.
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 31 | 31
units on a scale
  Baseline | 36.22 (12.32) | 38.05 (10.63)
  End of Treatment | 33.40 (9.15) | 34.12 (6.90)
  3-month followup | 29.80 (7.68) | 29.57 (6.31)

10. Secondary Outcome: Coping Skills Measure
Description: Self-report measure of confidence in ability to cope comprising 18 items, each scaled from 0 (not at all) to 5 (extremely). The mean across all 18 items ranges from 0 to 5 with higher scores indicating less pathology (i.e., stronger ability to cope).
Time Frame: Baseline, end of treatment, 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 31 | 31
units on a scale
  Baseline | 2.25 (1.09) | 2.92 (.40)
  End of Treatment | 2.88 (.99) | 2.95 (1.01)
  3-month followup | 2.85 (.69) | 2.92 (.40)

11. Secondary Outcome: Alcoholics Anonymous (AA) Intention Measure
Description: Self-reported attitudes toward attending 12-step meetings; a scale of 17 items, each rated 1 (extremely unlikely) to 7 (extremely likely). The mean across all items thus ranges from 1 to 7 with with more positive scores indicating a more positive attitude toward 12-step meetings.
Time Frame: Baseline, end of treatment (month 3), 3-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Number analyzed (Participants) | 29 | 28
units on a scale
  Baseline | 5.21 (1.27) | 5.26 (1.10)
  End of Treatment | 4.90 (1.42) | 4.97 (1.34)
  3-month followup | 4.99 (.98) | 4.97 (1.07)

ADVERSE EVENTS:
Time Frame: The full study period from each participant's randomization through 3-month followup.
Description: All serious adverse events reported were unrelated to the study and to the study treatments, as determined by our Institutional Review Board (IRB). Adverse events were monitored / reported only in terms of whether they were related or non-related to the study treatments, and not based on specific adverse event terms.
Arm/Group | A Woman's Path to Recovery (WPR) | 12-Step Facilitation (TSF)
Serious Adverse Events (participants affected / at risk) | 4/33 | 7/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Woman's Path to Recovery (WPR) (N=33) | 12-Step Facilitation (TSF) (N=33)
adverse events (Investigations) | 4 | 7 — All were determined to be unrelated to the study and study treatments, per the IRB of record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No